CLINICAL TRIAL: NCT01277068
Title: Effects of Various Bariatric Surgical Procedures on Intestinal Triglyceride-rich-lipoprotein (TRL) Metabolism in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2010-A00844-35
Record Dates: First submitted 2011-01-13; First posted 2011-01-14 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Obese Patients; Production Rates of These TRL Before and After the Bariatric Surgery; Cardiovascular Diseases
Keywords: obese patients; TRL; the bariatric surgery
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Surgical Procedures, Operative; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- the adjustable gastric banding (Active Comparator)
  Interventions: Procedure: Surgical and medical procedures
- the sleeve gastrectomy (Active Comparator)
  Interventions: Procedure: Surgical and medical procedures
- the gastric bypass (Active Comparator)
  Interventions: Procedure: Surgical and medical procedures

INTERVENTIONS:
Procedure: Surgical and medical procedures — this study want to compare the differential effect of the 3 bariatric surgery procedures on the production rates of the intestinal TRL: the adjustable gastric banding the sleeve gastrectomy the gastric bypass

SUMMARY:
Morbidly obesity (body mass index 40 kg/m²), the most serious, is more and more frequent. Cardiovascular diseases are the first cause of morbidity and mortality. An excess of TRL particles is one of the characteristics, represents a major cardiovascular risk factor. The overproduction of the intestinal TRL (which apoprotein B48 is the specific tracer) is recently recognized of insulin-resistance and the atherogenous role of these intestinal TRL has been shown. In front of this important overmortality, the bariatric surgery quickly developed. Three main procedures are performed: 2 based exclusively on the gastric restriction (the adjustable gastric banding and the sleeve gastrectomy) and one associating a malabsorption (the gastric bypass).

DETAILED DESCRIPTION:
It is a monocentric, prospective, comparative study. After identification of the eligible subjects, the kinetics (production and clearance rates) of the intestinal TRL will be performed in the hospital, using a stable isotope method (5,5,5-D3-L-Leucine), in 3 groups of obese patients (12 patients per surgery procedure), before and 6 months after the surgery

ELIGIBILITY:
Inclusion Criteria:

* Men or women from 18 to 65 years old
* Subject having a BMI included between 35 and 40 kg / m2 associated to at least a comorbidity susceptible to be improved after the surgery
* Subject in failure of a medical treatment, led by an expert in nutrition, associating a dietary coverage and a physical activity adapted for at least 6 months
* Subject without contraindication for 3 studied surgical techniques
* Subject without cardiovascular events 6 months ago
* subject is informed and is consented
* Subject having a biologic balance dating less than 3 months

Exclusion Criteria:

* subject with contraindication for 3 studied surgical techniques
* women pregnant
* subject did not consent and is not informed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2010-09; Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
to compare the differential effect of the 3 bariatric surgery procedures on the production rates of the intestinal TRL | 36 months
  the 3 bariatric surgery procedures are: the adjustable gastric banding the sleeve gastrectomy the gastric bypass (associating a malabsorption).

SECONDARY OUTCOMES:
to compare the production rates of these TRL before and after the bariatric surgery | 36 months
  TRL particles is one of the characteristics, represents a major cardiovascular risk factor. The overproduction of the intestinal TRL (which apoprotein B48 is the specific tracer) is a constituent recently recognized of insulin-resistance and the atherogenous role of these intestinal TRL has been shown

CONTACTS AND LOCATIONS:
Overall Officials: René Valero, Professor, Principal Investigator — APHM
Locations (1):
- Assistance Publique - Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Frances L, Croyal M, Ruidavets JB, Maraninchi M, Combes G, Raffin J, de Souto Barreto P, Ferrieres J, Blaak EE, Perret B, Moro C, Valero R, Martinez LO, Viguerie N. Identification of circulating apolipoprotein M as a new determinant of insulin sensitivity and relationship with adiponectin. Int J Obes (Lond). 2024 Jul;48(7):973-980. doi: 10.1038/s41366-024-01510-w. Epub 2024 Mar 15. PMID 38491190
- [Derived] Padilla N, Maraninchi M, Beliard S, Berthet B, Nogueira JP, Wolff E, Nicolay A, Begu A, Dubois N, Grangeot R, Mattei C, Vialettes B, Xiao C, Lewis GF, Valero R. Effects of bariatric surgery on hepatic and intestinal lipoprotein particle metabolism in obese, nondiabetic humans. Arterioscler Thromb Vasc Biol. 2014 Oct;34(10):2330-7. doi: 10.1161/ATVBAHA.114.303849. Epub 2014 Aug 7. PMID 25104797